CLINICAL TRIAL: NCT05509907
Title: Development of The Pediatric Physical Activity Tracking Platform (Pedi@Ctivity) and Smartwatch-based Big Data Analysis: A Digital Health Application in Society 5.0
Brief Title: Development of The Pediatric Physical Activity Tracking Platform (Pedi@Ctivity) and Smartwatch-based Big Data Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Nilay Arman, Assoc. Prof., Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 380972
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Physical Activity; Adolescent; Childhood Rheumatic Disease
Keywords: Physical Activity; Exercise; Big Data; Artificial Learning; Smart Watch; Adolescent; mHealth; ehealth
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy adolescents within 12-18 years old (Experimental): Adolescents aged 12-18 years who continue secondary education, do not have any chronic diseases or disabilities and volunteer to participate in the study will be included. Within the scope of the project, participants' demographic data, health parameters, physical fitness, functional capacity, fatigue level, exercise behavior, system availability and satisfaction will be evaluated. All evaluations, training on the use of smart watches and mobile and web-based physical activity tracking applications will be carried out at the school where the adolescents receive education.
  Interventions: Other: Pedi@ctivity Analysis and Tracking Mobile Applications and Web Platform
- Adolescents aged 12-18 years with chronic rheumatic disease (Experimental): Children with rheumatic disease who were diagnosed with chronic rheumatic disease, diagnosed at least 6 months ago, whose medical treatment was stable, and who volunteered to participate in the study will be included. Within the scope of the project, participants' demographic data, health parameters, physical fitness, functional capacity, fatigue level, exercise behavior, system availability and satisfaction will be evaluated. All assessments and training on smartwatches and mobile and web-based physical activity tracking applications will be held at Department of Pediatric Rheumatology, Istanbul Faculty of Medicine, Istanbul University.
  Interventions: Other: Pedi@ctivity Analysis and Tracking Mobile Applications and Web Platform

INTERVENTIONS:
Other: Pedi@ctivity Analysis and Tracking Mobile Applications and Web Platform — "Pedi@ctivity Analysis Mobile Application" and than Pedi@ctivity Analysis and Tracking Web Platform synchronized with the Pedi@ctivity Tracking Mobile Application, will be developed. The collected data will be analyzed with statistical methods and models using artificial intelligence algorithms will be created. According to the evaluations, physical activity and exercise videos and programs will be prepared and uploaded to web platform. Programs will include stretching, strengthening, balance, aerobic, calisthenic exercises and aerobic dance. The exercise and physical activity program will also be synchronized with the Pedi@ctivity Tracking Mobile Application and the smart watch. Pedi@ctivity Mobile Applications will provide health parameters from the smart watch, suggestions suitable for the exercise and physical activity program, and motivational feedback. Each adolescent will be included in a 3-month program. After the 3-month all evaluations at the beginning will be repeated.

SUMMARY:
Regular physical activity is extremely important for the protection and development of physical and psychosocial health. In addition, acquiring regular physical activity habits in the early years of life allows maintaining numerous gains related to physical fitness, functional capacity and psychoemotional health into adulthood.

Guided by scientific and technological innovations, focusing on sustainable development goals, the vision of Society 5.0 is based on digital innovation with artificial intelligence, the internet of things, digital technologies and big data, and is to increase the awareness of individuals and encourage individuals to take a role in improving their health status with wearable technology and mobile health applications. In the literature, only one study has been found on the acquisition of big data with wearable technologies for the promotion of physical activity in adolescents.

The general aim of our project is to obtain smartwatch-based big data for adolescents, which will be done for the first time in the field of health and sports in our country, and to analyze the obtained data using both statistical methods and big data analytics and artificial learning methods, to develop Pediatric Physical Activity Tracking Platform (Pedi@ktivite) through physical activity algorithms and to reveal the effect of the developed system on the physical fitness of adolescents and the usability of the system with scientific evidence. Within the scope of the project, adolescents with chronic rheumatic disease will also be included in the sample group, and the effects of the system to be developed in adolescents with the chronic rheumatic disease will be demonstrated. Due to the results obtained, we believe that this technology-supported approach will be an example of good practice for other chronic diseases.

As the first technology-supported and big data-oriented project for health and sports in adolescents, our project will fill an important gap and provide pioneering results for future projects, paving the way for providing services in the fields of health and sports with big data analytics and addressing physical inactivity.

ELIGIBILITY:
Inclusion Criteria:

* For Healthy Adolescent:

Adolescents aged 12-18 years who continue secondary education, Adolescents do not have any chronic diseases or disabilities Adolescents who volunteer to participate in the study

* Adolescents with chronic rheumatic disease:

Adolescents with rheumatism aged between 12-18 Adolescents with chronic rheumatic disease who volunteer to participate in the study

Exclusion Criteria:

* For Healthy Adolescent:

Adolescents who are older than 18 years of age, Adolescents who have had any discomfort or surgery that may affect their walking in the last 6 months, Adolescents and whose families are not asked to participate in the study

* Adolescents with chronic rheumatic disease:

Adolescents who are older than 18 years of age, Adolescents who have poor mental status, accompanying rheumatism and have additional neurological diagnosis that may affect the intervention results, Adolescents whose family does not want to participate in the study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Health Parameters | Change from Baseline Health Parameters at 12 weeks
  The adolescents included in the project will be given a smart watch and will be asked to use the watches for 3 months, and a training will be given to the adolescents on the use of smart watches by the project team. The data obtained on health-related parameters and physical activity behaviors of adolescents for 3 months through smart watches will be transferred to the cloud and web platform with the mobile application. With wearable activity tracker watches, data on the person's heart rate during the day, the number of steps taken per day, oxygen saturation, daily calories burned, activities performed and the locations where the activity is performed can be presented. There are many smart watches compatible with the Android OS operating system, it is planned to use 4 different smart watches in our project. With the mobile application we will develop in our project, the health parameters of adolescents using smart watches will be transferred to the platform.
FitnessGram Physical Activity Test Battery-Progressive Aerobic Cardiovascular Endurance Running (PACER) | Change from Baseline FitnessGram Physical Activity Test Battery-Progressive Aerobic Cardiovascular Endurance Running (PACER) at 12 weeks
  PACER is an adapted version of the 20 meter shuttle run test and is a field test consisting of multiple stages. The participant will run back and forth in a 20 meter area accompanied by the music coming from the voice recorder. The beep indicates when the participant should finish a lap. The test will start at slow speeds and will gradually increase each minute. The test will be terminated when the participant cannot continue to run at the level he has reached. The number of laps completed at the end of the test will be recorded. PACER is a more fun alternative to other distance running tests. It is recommended for use in children, adolescents and young adults. PACER will be used to assess the aerobic capacity of adolescents.
FitnessGram Physical Activity Test Battery-Bioelectrical Impedance Analysis | Change from Baseline FitnessGram Physical Activity Test Battery-Bioelectrical Impedance Analysis at 12 weeks
  BIA is based on the principle of measuring resistance to the flow of a low-level electric current through the body. In our study, body composition parameters such as muscle, fat and water ratio will be evaluated with the Tanita SC240 device.
FitnessGram Physical Activity Test Battery-Curl-up Test | Change from Baseline FitnessGram Physical Activity Test Battery-Curl-up Test at 12 weeks
  The participant will begin the test in the supine position, knees flexed approximately 140 degrees, feet flat on the floor, and legs slightly apart. The participant's arms will be parallel to the floor and torso. The palm will be positioned on the floor with the fingers stretched out. The purpose of this test is to do as many sit-ups as possible at a given speed. A maximum of 75 shuttles counts. The number of shuttles performed at the end of the test will be recorded. The curl-up test will be used to evaluate the abdominal muscle strength and endurance of adolescents.
FitnessGram Physical Activity Test Battery-Trunk Lift Test | Change from Baseline FitnessGram Physical Activity Test Battery-Trunk Lift Test at 12 weeks
  The participant will begin the test in the prone position with their hands placed under the thigh. A sign will be placed on the floor at the participant's eye level. During the movement, the participant will focus on this sign. During the test, the participant slowly and in a controlled manner raises their torso to a maximum height of 12 inches. The head is kept in neutral alignment with the spine. At the end of the test, the distance between the floor and the participant's chin will be measured with a ruler and the score will be recorded in centimeters (cm). Trunk lift test will be used to evaluate trunk extensor muscle strength and flexibility of adolescents.
FitnessGram Physical Activity Test Battery-Push-up Test | Change from Baseline FitnessGram Physical Activity Test Battery-Push-up Test at 12 weeks
  The participant will begin the test in the prone position, with their hands shoulder-width or wider than shoulder-width apart, fingers stretched, palms on the floor, and legs slightly apart. During the test, the participant lowers his torso towards the ground and raises himself up again when his elbows are bent 90º. The movement is repeated as much as possible. The rhythm is set to 20 push-ups per minute or 1 push-up per 3 seconds. The test is terminated when the participant makes a mistake twice. The number of push-ups performed at the end of the test will be recorded. The push-up test will be used to evaluate the upper extremity muscle strength and endurance of adolescents.
FitnessGram Physical Activity Test Battery-Back Saver Sit and Reach Test | Change from Baseline FitnessGram Physical Activity Test Battery-Back Saver Sit and Reach Test at 12 weeks
  During the test, the participant takes off his shoes and sits in front of the test apparatus. A box is needed for the test. This box is 35 cm long, 45 cm wide, 32 cm high. A top plate 55 cm long and 45 cm wide is put on top of the box. One leg of the participant is completely straight while the other is bent at the knee. The participant reaches forward four times with their hands on top of each other, holding the fourth reach position for 1 second. At the end of the test, the distance traveled will be recorded. The Back Saver Sit and Reach Test will be used to evaluate the hamstring flexibility of adolescents.
KFORCE Muscle Controller | Change from Baseline KFORCE Muscle Controller at 12 weeks
  The KFORCE Muscle Controller is a handheld dynamometer for the evaluation of muscle strength. It assesses maximum strength, endurance, and muscle symmetry. The Muscle controller is versatile and adaptable to many configurations. As a result of the evaluation, the participant's results are recorded in a database. Then, the progress of the participant can be followed in the database of the application. Muscle strength of adolescents will be evaluated with the device.
KFORCE Plates | Change from Baseline KFORCE Plates at 12 weeks
  KFORCE Plates is a strength platform used to improve balance and assess lower extremity muscle symmetry and strength. It consists of two independent plates. KFORCE plates allow the measurement of static and dynamic balance in a wide range of movements. In addition, it can determine the center of gravity and measure the weight distribution in the stance phase. It evaluates squatting, push-ups and jumping characteristics and presents a report containing multiple data as a result of the measurement. Static and dynamic balance analyzes of adolescents will be made with the device.
KFORCE Sens | Change from Baseline KFORCE Sens at 12 weeks
  KFORCE Sens is an electronically linked goniometer. It allows the evaluation and monitoring of the range of motion of the body joints. With KFORCE Sens, the maximum amplitude of motion can be measured for a specific body joint in a specific anatomical plane. The dynamic balance of adolescents during running and walking will be evaluated with the system. Adolescents' joint range of motion will be evaluated with KFORCE Sens.
Smart Insole PODOSmart (Digitsole) | Change from Baseline Smart Insole PODOSmart (Digitsole) at 12 weeks
  PODOSmart®insoles consists of wireless sensors, can be fitted intoany shoe and offer the ability to measure spatial, temporal, and kinematic gait parameters. The intelligent insoles feature several sensors that detect and capture foot movements and a microprocessorthat calculates gait related biomechanical data. Each PODOSmart®insole has an inertial platform that records each foot's walking steps, running strides, and orientations in space with sampling frequency of 208 Hz for walk analysis.The Bluetooth connection box retrieves the collected data by the smart insoles. Then,those data are processed by proprietary artificial intelligence algorithms to calculate thespatiotemporal, kinematic, and biomechanical parameters.The dynamic balance of adolescents during running and walking will be evaluated with the system.
6 Minute Walk Test (6 MWT) | Change from Baseline 6 Minute Walk Test (6 MWT) at 12 weeks
  The 6-minute walk test is a well-tolerated, easy-to-apply and simple test that shows the submaximal level of functional capacity. This test measures the distance that participants can walk quickly on a hard and flat surface in 6 minutes. Participants rest in a chair near the starting position for at least 10 minutes before the start of the test. Before and after the test, heart rate, blood pressure, saturation are measured, and fatigue level is determined with the Modified Borg scale. Participants are told how to perform the test. At the end of the test, the distance walked by the participants in 6 minutes will be recorded in meters. The 6 Minute Walk Test will be used to evaluate the functional capacities of adolescents.
Visual Analogue Scale (VAS) | Change from Baseline Visual Analogue Scale (VAS) at 12 weeks
  A 100 millimeter (mm) VAS will be used to assess the fatigue severity of the participants. According to the VAS, scores <20 mm mean "low fatigue", scores between 20-49 mm mean "clinically significant fatigue" and scores ≥50 mm mean "severe fatigue".
Exercise Stage of Change Scale Short Form | Change from Baseline Exercise Stage of Change Scale Short Form at 12 weeks
  "Exercise Exercise Stage of Change Scale Short Form" consists of five questions. The participant is asked to choose only one of the five situations that fit the current exercise level. These questions reveal the stage of change that the individual is in.
Decisional Balance Scale in Exercise | Change from Baseline Decisional Balance Scale in Exercise at 12 weeks
  It evaluates the individual's subjective perception of the perceived benefits of exercising and the perceived harms of not exercising, which have an effect on the individual's exercise behavior. In the scale consisting of 10 items. Regarding the decision to exercise or not to exercise in their spare time, why each situation is important for individuals is determined using a 5-point Likert scale. The total score of the scale is obtained by subtracting the total score of perceived harm from the total score of perceived benefit of exercise.The highest score that can be obtained from the scale is 25, and the lowest score is 5.The perception of the subjects to exercise will be evaluated with the "Decisional Balance Scale in Exercise".
System Usability Scale | Change from Baseline System Usability Scale at 12 weeks
  Detectability and usability of interactive systems will be evaluated with the "System Usability Scale". It is a scale consisting of 10 questions commonly used in the literature. It is scored from 1 (strongly disagree) to 5 (strongly agree). A high total score indicates that the system is detectable and usable.
Numerical Rating Scale | Change from Baseline Numerical Rating Scale at 12 weeks
  Children's satisfaction with the use of physical activity tracking platform and smart watch will be evaluated with the "Numerical Rating Scale" with 0-10 points. A high score indicates a high level of satisfaction. Children's satisfaction level with the system will be evaluated with the "Numerical Rating Scale".

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, Assoc.Prof., Principal Investigator — Istanbul University-Cerrahpaşa, Faculty of Health Science, Department of Physiotherapy and Rehabilitation; Asya Albayrak, Pt., MSc., Study Chair — Istanbul University-Cerrahpasa, Institute of Postgraduate Education; Asena Yekdaneh, Pt., MSc., Study Chair — Istanbul University-Cerrahpasa, Institute of Postgraduate Education; Tuna Cakar, Assist. Prof., Study Chair — MEF University, Department of Computer Engineering; Nuray Aktay Ayaz, Prof. Dr., Study Chair — Istanbul Faculty of Medicine, Department of Internal Medicine, Department of Pediatric Rheumatology; Sevim Gullu, Assoc. Prof., Study Chair — Istanbul University-Cerrahpasa, Faculty of Sports Sciences, Department of Recreation; Alperen Sayar, Study Chair — MEF University, Graduate School of Science and Engineering,Department of Information Technologies; Tunahan Bozkan, Study Chair — MEF University, Graduate School of Science and Engineering,Department of Information Technologies
Locations (1):
- İstanbul Tıp Fakültesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No